CLINICAL TRIAL: NCT01892007
Title: Evaluation of Cogmed Working Memory Training to Improve Cognition, Speech Perception and Self-reported Hearing Abilities for Adult Hearing Aid Users: a Double-blind, Randomised, Active-controlled Trial.
Brief Title: Evaluation of Cogmed Working Memory Training for Adult Hearing Aid Users
Acronym: TEACH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08ET002-01
Record Dates: First submitted 2013-06-27; First posted 2013-07-03 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Hearing Loss
Keywords: Hearing loss; Hearing aid; Speech intelligibility; Speech perception; Cognitive training; Working memory; Working memory training
MeSH Terms: conditions — Hearing Loss; Speech Intelligibility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cogmed RM (adaptive) (Experimental): Online training intervention: An adaptive version of Cogmed RM working memory training. Task difficulty (number of to-be-remembered items) increases based on individual performance, in order to maintain average daily performance levels of approximately 60% of trials correct. Participants complete 35-45 minutes of active training per day, 5 days a week for 5 weeks.
  Interventions: Behavioral: Cogmed RM - Online adaptive working memory training
- Cogmed RM (non-adaptive, placebo) (Placebo Comparator): Online training intervention: A non-adaptive placebo version of Cogmed RM working memory training. Tasks are fixed at a low-difficulty practice level (three to-be-remembered items) and do not increase in difficulty over the course of the intervention. Participants complete 35-45 minutes of active placebo training per day, 5 days a week for 5 weeks.
  Interventions: Behavioral: Cogmed RM - Online non-adaptive (placebo) working memory training

INTERVENTIONS:
Behavioral: Cogmed RM - Online adaptive working memory training
  Arms: Cogmed RM (adaptive)
Behavioral: Cogmed RM - Online non-adaptive (placebo) working memory training
  Arms: Cogmed RM (non-adaptive, placebo)

SUMMARY:
A double-blind randomised active-controlled trial aims to assess whether Cogmed (adaptive) working memory training results in improvements in untrained measures of cognition, speech perception and self-reported hearing abilities in older adults (50-74 years) with mild-moderate hearing loss who are existing hearing aid users, compared with an active placebo Cogmed (non-adaptive) control. It is hypothesised that improvements on trained Cogmed tasks, representing increased working memory capacity, will result in improved performance on cognitive and speech perception tasks that engage working memory. We also measure self-reported hearing ability to assess self-perceived benefit of Cogmed training.

DETAILED DESCRIPTION:
One in ten people aged between 55-74 years have a significant hearing impairment in their better hearing ear (as defined by audiometric hearing thresholds). Yet, it is becoming increasingly clear that the challenges faced by older listeners cannot be explained by the audiogram. The ability for people with hearing loss to use cognition to support context allows for compensation of degraded auditory input, which in turn offers promise for new cognitive-based rehabilitative interventions. Working memory is known to be highly associated with language and recent evidence has shown significant generalisation of on-task learning from Cogmed working memory training to improvements in sentence-repetition skills of children with severe to profound hearing loss and use cochlear implants. This evidence offers support for further investigation into the potential benefits of working memory training to improve speech perception abilities in other hearing impaired populations. This study aims to assess whether Cogmed (adaptive) working memory training improves the listening abilities of adults with mild to moderate hearing loss as assessed using untrained measurers of cognition, speech perception and self-reported hearing ability, compared with an active control (Cogmed, non-adaptive) group. A 6 month follow-up will assess retention of any training-related improvements in outcomes for the adaptive training group.

ELIGIBILITY:
Inclusion criteria:

* Existing (3+ months) hearing aid(s) user
* Mild to moderate (PTA0.25-4k Hz 21-69 dB HL) sensorineural hearing loss (SNHL) in the better hearing ear (SNHL defined as air-bone gap across 0.5k, 1k & 2k Hz < 15 dB)
* Internet access at home

Exclusion criteria:

* Participation in a previous training intervention study
* First language other than English (all speech outcome measure are presented in English)
* Unable to use either a desktop or laptop computer (Cogmed RM working memory training is delivered via the internet using a desktop or laptop computer)
* Cognitive impairment as defined as a score of less than 26/30 (fail) on the Montreal Cognitive Assessment (MoCA)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Henshaw, PhD, Principal Investigator — NIHR Nottingham Hearing Biomedical Research Unit, University of Nottingham.; Melanie Ferguson, BSc (Hons), Study Director — NIHR Nottingham Hearing Biomedical Research Unit, University of Nottingham.
Locations (1):
- QMC Ropewalk House, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Henshaw H, Heinrich A, Tittle A, Ferguson M. Cogmed Training Does Not Generalize to Real-World Benefits for Adult Hearing Aid Users: Results of a Blinded, Active-Controlled Randomized Trial. Ear Hear. 2022 May/Jun;43(3):741-763. doi: 10.1097/AUD.0000000000001096. PMID 34524150
- [Derived] Henshaw H, Ferguson MA. Working memory training for adult hearing aid users: study protocol for a double-blind randomized active controlled trial. Trials. 2013 Dec 5;14:417. doi: 10.1186/1745-6215-14-417. PMID 24304745

RESULTS

PARTICIPANT FLOW:
Groups:
- Cogmed RM (Adaptive): Online training intervention: An adaptive version of Cogmed RM working memory training. Task difficulty (number of to-be-remembered items) increases based on individual performance, in order to maintain average daily performance levels of approximately 60% of trials correct. Participants complete 35-45 minutes of active training per day, 5 days a week for 5 weeks.
  Cogmed RM - Online adaptive working memory training intervention
- Active Control: Cogmed RM (Non-adaptive, Placebo): Online training intervention: A non-adaptive placebo version of Cogmed RM working memory training. Tasks are fixed at a low-difficulty practice level (three to-be-remembered items) and do not increase in difficulty over the course of the intervention. Participants complete 35-45 minutes of active placebo training per day, 5 days a week for 5 weeks.
  Cogmed RM - Online (non-adaptive, placebo) working memory training intervention
Period: Overall Study
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Started | 27 | 30
Completed | 27 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo) | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.3) | 63.7 (5.5) | 64.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 13 | 14 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27 | 30 | 57
Montreal Cognitive Assessment (MoCA) score [Mean (Standard Deviation); unit: MoCA score] — Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal cognitive functioning.
  MoCA score | 27.9 (1.2) | 28.1 (1.6) | 28.0 (1.4)
BE PTA (0.25-4k Hz) [Mean (Standard Deviation); unit: decibels] — Better ear pure tone audiometric thresholds measured in decibels (dB) averaged across octave frequencies 0.25, 0.5, 1k, 2k and 4k Hz.
  On the decibel scale, the quietest audible sound (perceived near total silence) is 0 dB. A sound 10 times more powerful is 10 dB. Lower pure-tone audiometric thresholds indicate better hearing.
  decibels | 43.3 (14.5) | 37.5 (12.5) | 40.2 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Visual Letter Monitoring Task
Description: The VLM is a visual task of working memory (Gatehouse, Naylor, & Elberling, 2006) that is not trained within the Cogmed working memory training program. Ten consonant-vowel-consonant (CVC) words are embedded in an 80-letter sequence. Two sequences are presented to participants at each outcome assessment in a counterbalanced order. Individual letters are displayed sequentially on a computer screen at a rate of 2 second per letter (first list) and 1 second per letter (second list). Participants were asked to press the keyboard 'space bar' (hit) when three consecutive letters formed a recognised CVC word (for example, M-A-T). Task performance was scored as the total number of hits (maximum score of ten per list). Higher scores indicate better performance.
Time Frame: 0, 2, 7, and (adaptive training group only) 31 weeks
Population: Outcome measured at 0, 2, 7 and (adaptive training group only) 31 weeks. Training-related improvements in outcomes are assessed using the change in performance between pre-training (2 weeks) to post-training (7 weeks) measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
score on a scale
  (VLM 2 second) 0 weeks | 8.48 (1.42) | 8.27 (1.89)
  (VLM 2 second) 2 weeks | 8.07 (2.59) | 8.73 (1.48)
  (VLM 2 second) 7 weeks | 8.33 (2.04) | 8.93 (1.55)
  (VLM 2 second) 31 weeks: number analyzed (Participants) | 27 | 0
  (VLM 2 second) 31 weeks | 8.63 (1.97) |
  (VLM 1 second) 0 weeks | 5.74 (2.36) | 6.67 (2.50)
  (VLM 1 second) 2 weeks | 5.93 (2.95) | 6.93 (2.56)
  (VLM 1 second) 7 weeks | 6.73 (2.01) | 7.07 (2.73)
  (VLM 1 second) 31 weeks: number analyzed (Participants) | 27 | 0
  (VLM 1 second) 31 weeks | 6.50 (2.25) |

2. Secondary Outcome: Phonemic Discrimination Probe
Description: The phoneme discrimination task assesses an individual's ability to distinguish differences between phonemes presented on a continuum. Participants were presented with three discrete phonemes per trial from a continuum of 96 sound files (48 for each phoneme within a pair). For each trial, two of the phonemes were identical and one was different. Participants were asked to identify the odd one out. Two different phoneme pairs: /a/ /e/ (easy) and /d/ /g/ (difficult) were presented for a block of 35 trials in sequential blocks, with a 3-trial demonstration of continuum /a/ /e/. The task was presented in quiet room and difficulty was adapted based on individual participant performance using a three-phase adaptive staircase procedure (Moore, 2005) to provide a phoneme discrimination threshold, which is calculated as the average distance between the 96 sound files for the last 2 reversals in a block of 35 trials. Scores range from 50-100, with lower scores indicating better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
score on a scale
  (PD /e/ /a/) 0 weeks | 69.98 (8.97) | 73.79 (13.58)
  (PD /e/ /a/) 2 weeks | 65.92 (7.39) | 68.47 (11.93)
  (PD /e/ /a/) 7 weeks | 69.59 (11.67) | 65.20 (9.58)
  (PD /e/ /a/) 31 weeks: number analyzed (Participants) | 27 | 0
  (PD /e/ /a/) 31 weeks | 64.96 (8.39) |
  (PD /d/ /g/) 0 weeks | 86.44 (11.26) | 89.88 (10.18)
  (PD /d/ /g/) 2 weeks | 89.10 (11.46) | 87.07 (12.65)
  (PD /d/ /g/) 7 weeks | 90.07 (11.00) | 88.40 (12.09)
  (PD /d/ /g/) 31 weeks: number analyzed (Participants) | 27 | 0
  (PD /d/ /g/) 31 weeks | 85.67 (13.63) |

3. Secondary Outcome: BESST High/Low Context Sentence Intelligibility
Description: Based on the Revised Speech Perception in Noise Test (Bilger et al, 1984; Kalikow et al, 1977), the British English Semantic Sentence Test (BESST) stimuli are produced by a British English native speaker. Lists of 22 sentences (11 high-predictability and 11 low-predictability) were presented in the freefield in a background of speech-modulated noise with the same long-term average spectrum as the target speech (Knight, 2017), at a fixed signal-to-noise ratio (SNR) of -1 decibel (dB) SNR. Two practice sentences (one high- and one low-predictability) were presented to participants at a slightly more favourable fixed SNR (2 dB SNR) prior to commencing the main test. Participants were asked to listen to each sentence and repeat the last word aloud. The task was scored as the percentage of last words correctly repeated for both high-predictability and low-predictability lists. Higher scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of last words correct
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
percentage of last words correct
  BESST (High Context) 0 weeks | 31.65 (23.92) | 33.23 (26.07)
  BESST (High Context) 2 weeks | 30.18 (18.47) | 24.16 (17.90)
  BESST (High Context) 7 weeks | 29.98 (23.22) | 29.48 (21.12)
  BESST (High Context) 31 weeks: number analyzed (Participants) | 27 | 0
  BESST (High Context) 31 weeks | 22.73 (21.77) |
  BESST (Low Context) 0 weeks | 15.65 (14.51) | 14.75 (13.19)
  BESST (Low Context) 2 weeks | 21.10 (16.33) | 22.90 (14.09)
  BESST (Low Context) 7 weeks | 18.20 (16.73) | 18.20 (13.53)
  BESST (Low Context) 31 weeks: number analyzed (Participants) | 27 | 0
  BESST (Low Context) 31 weeks | 18.66 (14.61) |

4. Secondary Outcome: Modified Coordinate Response Measure (MCRM)
Description: The MCRM is a measure of target talker speech perception in the presence of another talker, presented at an adaptive signal-to-noise ratio (SNR). Participants were presented with sentences in the form of 'show the [animal] where the [color] [number] is'. Participants were asked to listen for the color and number spoken by the female speaker ('dog' was always the animal target) while ignoring the male speaker, and respond by pressing the corresponding target color number on a touchscreen computer. The test used an adaptive 1-up 1-down staircase method and continued until a total of eight reversals were achieved. The test was completed twice by each participant and a third time for instances where there was a difference of ≥5 decibel (dB) SNR between participants' first two test scores. Speech reception thresholds were calculated using the average of the last two reversals, averaged across the 2 or 3 tests. Lower scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
decibels
  MCRM 0 weeks | -3.88 (4.85) | -5.15 (5.68)
  MCRM 2 weeks | -4.51 (5.66) | -6.50 (5.66)
  MCRM 7 weeks | -4.69 (5.40) | -6.76 (5.01)
  MCRM 31 weeks: number analyzed (Participants) | 27 | 0
  MCRM 31 weeks | -4.05 (4.79) |

5. Secondary Outcome: Digit Span Backwards
Description: A subtest from the Wechsler Adult Intelligence Scale, Third Edition (WAIS-III) (Wechsler, 1997), this task involved listening to a string of numbers of increasing length and repeating them in reverse order. The test was presented using pre-recorded digits delivered using the Medical Research Council (MRC) Institute of Hearing Research System for Testing Auditory Responses (IHR-STAR) platform via a speaker situated directly in front of the participant. Trials began with strings of two numbers, finishing at strings of eight. Each string length was presented twice. Strings increased in length by one digit if participants correctly recalled one of the two digit strings at each length, otherwise the test was discontinued. Task performance was scored as the total number of strings correctly recalled in reverse order (of a maximum 14 trials). Higher scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: trials correct
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
trials correct
  Digit Span (BW) 0 weeks | 6.96 (2.10) | 7.17 (2.83)
  Digit Span (BW) 2 weeks | 7.69 (1.78) | 8.00 (3.06)
  Digit Span (BW) 7 weeks | 8.76 (2.19) | 7.83 (2.67)
  Digit Span (BW) 31 weeks: number analyzed (Participants) | 27 | 0
  Digit Span (BW) 31 weeks | 8.82 (2.36) |

6. Secondary Outcome: Test of Attention in Listening (TAIL)
Description: The Test of Attention in Listening (TAIL) is a measure of auditory attention using tones that vary in both frequency and spatial location (Zhang et al., 2012). Primary tasks included both frequency and location discrimination and participants were asked to respond as to whether two tones were the 'same' or 'different' in terms of either frequency or location . Tones were presented in the freefield at participants' most comfortable loudness (MCL) level (Ventry et al., 1971) via two speakers situated at 90° to the left and 90° to the right of the participant at a distance of 50cm. TAIL measures the ability to focus selectively on a task-relevant dimension (either frequency or location) and ignore information from task-irrelevant dimensions, using reaction time (RT) as the primary performance measure. This test produced two measures per condition (frequency and location), calculated from the RT data; Distraction and Conflict Resolution. Lower scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
seconds
  TAIL (Attend Frequency_Distraction) 0 weeks | 0.056 (0.145) | 0.038 (0.108)
  TAIL (Attend Frequency_Distraction) 2 weeks | 0.013 (0.130) | 0.074 (0.131)
  TAIL (Attend Frequency_Distraction) 7 weeks | 0.033 (0.144) | 0.056 (0.100)
  TAIL (Attend Frequency_Distraction) 31 weeks: number analyzed (Participants) | 27 | 0
  TAIL (Attend Frequency_Distraction) 31 weeks | 0.064 (0.108) |
  TAIL (Attend Frequency_Conflict Res) 0 weeks | -0.023 (0.089) | -0.023 (0.115)
  TAIL (Attend Frequency_Conflict Res) 2 weeks | 0.017 (0.109) | 0.047 (0.105)
  TAIL (Attend Frequency_Conflict Res) 7 weeks | 0.006 (0.105) | 0.051 (0.125)
  TAIL (Attend Frequency_Conflict Res) 31 weeks: number analyzed (Participants) | 27 | 0
  TAIL (Attend Frequency_Conflict Res) 31 weeks | 0.047 (0.091) |
  TAIL (Attend Location_Distraction) 0 weeks | 0.108 (0.110) | 0.108 (0.133)
  TAIL (Attend Location_Distraction) 2 weeks | 0.108 (0.126) | 0.082 (0.115)
  TAIL (Attend Location_Distraction) 7 weeks | 0.097 (0.140) | 0.094 (0.097)
  TAIL (Attend Location_Distraction) 31 weeks: number analyzed (Participants) | 27 | 0
  TAIL (Attend Location_Distraction) 31 weeks | 0.119 (0.150) |
  TAIL (Attend Location_Conflict Res) 0 weeks | 0.1097 (0.125) | 0.095 (0.147)
  TAIL (Attend Location_Conflict Res) 2 weeks | 0.105 (0.134) | 0.095 (0.098)
  TAIL (Attend Location_Conflict Res) 7 weeks | 0.136 (0.119) | 0.099 (0.081)
  TAIL (Attend Location_Conflict Res) 31 weeks: number analyzed (Participants) | 27 | 0
  TAIL (Attend Location_Conflict Res) 31 weeks | 0.155 (0.168) |

7. Secondary Outcome: Test of Everyday Attention Subtests 6 & 7
Description: The Test of Everyday Attention (TEA) subtests 6 (telephone search) and 7 (telephone search while counting) assess single (visual) attention and dual (auditory and visual) attention (Robertson, Ward, Ridgeway, & Nimmo-Smith, 1994). For subtest 6, participants were asked to search a telephone directory for matching symbols. For subtest 7, participants were asked to search a telephone directory for matching symbols while counting strings of beeps in varying lengths (2 to 12) presented in the freefield. The task as scored using time (seconds) per correctly identified symbol, weighted in subtest 7 by the proportion of correctly counted beep strings. A dual task decrement was calculated as the difference in time (in seconds) per correctly identified symbol where two simultaneous tasks are being completed, compared with that for a single task (subtest 7 minus subtest 6). Lower scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
seconds
  (TEA 6) 0 weeks | 4.11 (3.67) | 3.35 (0.65)
  (TEA 6) 2 weeks | 3.27 (0.63) | 3.23 (0.70)
  (TEA 6) 7 weeks | 3.25 (0.66) | 3.00 (0.69)
  (TEA 6) 31 weeks: number analyzed (Participants) | 27 | 0
  (TEA 6) 31 weeks | 3.09 (0.55) |
  (TEA 7) 0 weeks | 0.12 (3.03) | 1.26 (1.48)
  (TEA 7) 2 weeks | 1.11 (1.95) | 1.26 (2.98)
  (TEA 7) 7 weeks | 0.80 (1.06) | 0.55 (0.78)
  (TEA 7) 31 weeks: number analyzed (Participants) | 27 | 0
  (TEA 7) 31 weeks | 0.81 (0.92) |

8. Secondary Outcome: Size Comparison Span
Description: The size-comparison span (SICSPAN) task (Sorqvist, Ljungberg, & Ljung, 2010) asked participants to view lists of size comparisons (e.g. 'tree is larger than acorn') and respond 'yes' or 'no' using a button box. Participants were then provided with to-be-remembered words from the same semantic category (e.g. 'leaf'). At the end of the list, participants were required to recall the to-be-remembered words while inhibiting words included in the size comparison judgments. The task began with lists of 2 size comparison judgments and to-be-remembered words, increasing to list lengths of 3, 4, 5 and 6. There were two trials at each list length. The task continued until all list lengths had been presented, with no discontinuation rule. The task was scored using the number of list items correctly recalled (maximum 40). A second measure (intrusions) recorded the number of incorrect items recalled, or errors in inhibition, for each participant. Higher scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
score on a scale
  SICSPAN (total) 0 weeks | 20.96 (6.16) | 24.40 (7.82)
  SICSPAN (total) 2 weeks | 24.26 (7.02) | 26.27 (8.31)
  SICSPAN (total) 7 weeks | 25.11 (7.05) | 26.43 (8.16)
  SICSPAN (total) 31 weeks: number analyzed (Participants) | 27 | 0
  SICSPAN (total) 31 weeks | 24.64 (6.07) |
  SICSPAN (intrusions) 0 weeks | 4.82 (3.63) | 3.20 (2.33)
  SICSPAN (intrusions) 2 weeks | 5.11 (4.10) | 3.97 (3.35)
  SICSPAN (intrusions) 7 weeks | 4.52 (4.01) | 410 (3.68)
  SICSPAN (intrusions) 31 weeks: number analyzed (Participants) | 27 | 0
  SICSPAN (intrusions) 31 weeks | 5.59 (4.15) |

9. Secondary Outcome: Dual Task of Listening and Working Memory
Description: The dual task is a measure of listening and memory designed to assess listening effort (Howard, Munro, & Plack, 2010). Participants were presented with a 5-digit memory task that flanked a speech-in-noise comprehension task. A string of 5 digits was displayed visually on a computer screen for 5 seconds. Participants were asked to retain the digits in memory for later recall. Participants were then presented with a list of 5 Arthur Boothroyd (AB) isophonemic monosyllabic words (Boothroyd, 1968) presented in multi-talker babble, and were asked to repeat each word immediately after presentation. After each list of five words, participants were asked to recall the previously presented five digits. There were 4 word lists, resulting in a maximum possible score of 20 correctly repeated words and 20 correctly recalled digits. A dual-task score was calculated by adding together the scores for the word and digit tasks (maximum 40). Higher scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
score on a scale
  Dual Task 0 weeks | 18.11 (6.66) | 18.87 (5.14)
  Dual Task 2 weeks | 19.26 (5.77) | 20.20 (6.20)
  Dual Task 7 weeks | 20.88 (5.73) | 22.14 (5.53)
  Dual Task 31 weeks: number analyzed (Participants) | 27 | 0
  Dual Task 31 weeks | 20.71 (5.14) |

10. Secondary Outcome: Hearing Handicap Inventory for the Elderly (HHIE)
Description: The Hearing Handicap Inventory for the Elderly is a 25-item validated questionnaire that quantifies the emotional and social/situational effects of self-perceived hearing impairment to quantify hearing-specific quality of life. Participants were asked to complete the 25-item paper questionnaire answering statements such as 'Does a hearing problem cause you to be nervous' with either 'yes' (4 points), 'no' (0 points) or 'sometimes' (2 points). The questionnaire was scored as total points for all items (maximum 100 points). Subtotal scores can also be derived for emotional (12 items, maximum 48 points) and situational item subscales (13 items, maximum 52 points). Lower scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
score on a scale
  HHIE 0 weeks | 40.89 (27.10) | 34.07 (21.36)
  HHIE 2 weeks | 39.93 (27.90) | 30.73 (23.75)
  HHIE 7 weeks | 37.19 (26.84) | 28.41 (21.19)
  HHIE 31 weeks: number analyzed (Participants) | 27 | 0
  HHIE 31 weeks | 35.90 (30.04) |

11. Secondary Outcome: Glasgow Hearing Aid Benefit Profile (GHABP)
Description: The Glasgow Hearing Aid Benefit Profile (GHABP) is a validated questionnaire to assess self-reported activity limitations (GHABP Initial Disability) and participation restrictions (GHABP Handicap) arising from difficulties in hearing, as well as hearing aid use, benefit, and satisfaction (Gatehouse, 1999). For the purposes of the present study population (experienced hearing aid users) only the first two measures were assessed. Participants were presented with four listening scenarios and were asked to rate the amount of difficulty they have in that situation while wearing their hearing aids (1 = no difficulty to 5 = cannot manage at all), together with how much any difficulty either worried, annoyed or upset them ( 1 = not at all to 5 = very much indeed). The mean of all four scenarios in each measure were converted to a percentage score for GHABP Initial Disability and GHAPB Handicap. Lower scores indicate better performance.
Time Frame: 0, 2, 7 and (adaptive training group only) 31 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
Number analyzed (Participants) | 27 | 30
units on a scale
  GHABP (Initial Disability) 0 weeks | 43.29 (16.98) | 35.00 (15.54)
  GHABP (Initial Disability) 2 weeks | 43.98 (17.80) | 36.42 (15.68)
  GHABP (Initial Disability) 7 weeks | 38.66 (20.07) | 36.88 (15.77)
  GHABP (Initial Disability) 31 weeks: number analyzed (Participants) | 27 | 0
  GHABP (Initial Disability) 31 weeks | 36.84 (22.77) |
  GHABP (Handicap) 0 weeks | 35.88 (26.21) | 29.38 (19.91)
  GHABP (Handicap) 2 weeks | 34.26 (28.82) | 29.31 (20.46)
  GHABP (Handicap) 7 weeks | 30.56 (29.89) | 24.38 (16.93)
  GHABP (Handicap) 31 weeks: number analyzed (Participants) | 27 | 0
  GHABP (Handicap) 31 weeks | 30.40 (28.56) |

ADVERSE EVENTS:
Arm/Group | Cogmed RM (Adaptive) | Active Control: Cogmed RM (Non-adaptive, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No